CLINICAL TRIAL: NCT00945867
Title: The Use of CYP 450 2D6 Genotype as a Predictor of Flecainide Efficacy in the Treatment of Patients With Atrial Fibrillation
Brief Title: Cytochrome P450 2D6 (CYP 450 2D6) Genotype and Flecainide Efficacy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Therese Fuchs, MD, Assaf Harofeh Medical Center
Other Study IDs: 111/09
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2009-07

CONDITIONS: Atrial Fibrillation
Keywords: flecainide; pharmacogenetics
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The determination of the 2D6 genotype will enable us to determine the way flecainide is metabolized by the liver. Some individuals are poor metabolizers and some individuals are extensive metabolizers of the drug. This will also determine which patients will benefit from the drug.

DETAILED DESCRIPTION:
Pharmacogenetics is the study of genetic variations on drug metabolizing enzymes and transporters. Pharmacogenetics is one of the first clinical applications of the Human Genome Project. Pharmacogenomics is the study of the role of interindividual genomics variability on drug response, efficacy, and metabolism. It correlates the effects of the entire expressed genome to the clinical usefulness and toxicity of a drug. Pharmacogenomics has the potential to change the way patients' therapy is optimized, allowing an era of "personalized medicine" in which patients will be divided into groups based on genetic markers that treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent AF
* Patients with a structurally normal heart
* Patients > 18 YO
* Patients who signed an informed consent

Exclusion Criteria:

* Renal failure with creatinine clearance less than 40
* Elevated liver enzymes 3 times the normal range, or causing coagulation test abnormality
* Pregnant patients
* Patients treated with psychiatric agents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation and a normal heart.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
no recurrence of atrial fibrillation | 3 months

SECONDARY OUTCOMES:
the dose of flecainide used | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Sharist, MD, Study Chair — Assaf-Harofeh Medical Center; Shmuel Bar-Haim, MD, Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Zrifin, Israel